CLINICAL TRIAL: NCT04557176
Title: TB Screening Improves Preventive Therapy Uptake Trial
Brief Title: TB Screening Improves Preventive Therapy Uptake
Acronym: TB SCRIPT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Makerere University (Other); Infectious Diseases Research Collaboration, Uganda (Other); Johns Hopkins University (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: 18-25623; 1R61HL146365-01A1 (NIH)
Record Dates: First submitted 2020-09-14; First posted 2020-09-21 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Tuberculosis; Latent Tuberculosis; Tuberculosis Prevention; HIV
Keywords: Tuberculosis; Latent tuberculosis; Tuberculosis preventive therapy; HIV; C-reactive protein; Symptom screening; Intensified case finding
MeSH Terms: conditions — Tuberculosis; Latent Tuberculosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Masking will be maintained by administering finger prick tests to all participants, irrespective of trial arm. Intervention arm participants will have CRP levels measured from blood obtained by finger prick. Control arm participants will have beta-human chorionic gonadotropin (beta-hCG) levels measured from blood obtained by finger prick.
  Only participants, study investigators and routine clinical care providers will be masked. Study staff performing TB screening in accordance with the participant's randomization assignment and activities downstream of TB screening (i.e., confirmatory TB testing, TPT eligibility assessment) will not be masked. The database administrator will have access to the randomized assignments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- POC CRP-based TB screening (Experimental): Participants randomized to the intervention arm will undergo POC CRP-based TB screening at study entry. Participants with elevated POC CRP levels (≥8 mg/L) will be regarded as screen-positive and will be referred for confirmatory TB testing. Participants with non-elevated POC CRP levels (<8 mg/L) will be regarded as screen-negative and will be assessed for TPT eligibility.
  Interventions: Device: CRP, point-of-care assay
- Symptom-based TB screening (No Intervention): Participants randomized to the control arm will undergo symptom-based TB screening at study entry. Participants reporting ≥1 TB symptom (current cough, fever, night sweats, weight loss) will be regarded as screen-positive and will be referred for confirmatory TB testing, in accordance with WHO guidelines. Participants with none of the 4 TB symptoms will be regarded as screen-negative and will be assessed for TPT eligibility.

INTERVENTIONS:
Device: CRP, point-of-care assay — CRP is a non-specific marker of inflammation whose levels rise in the setting of interleukin 6 (IL-6)-mediated inflammation, such as active TB. In clinical settings, CRP is used to identify patients with systemic inflammation from infection or non-infectious cases. In settings with high TB prevalence, the investigators hypothesize that CRP can be used to accurately screen individuals for active TB (i.e., distinguish individuals with high likelihood of having active TB from those individuals unlikely to have active TB).
  Other Names: iCHROMA CRP reader; Boditech Med Inc.
  Arms: POC CRP-based TB screening

SUMMARY:
HIV-infected people have an increased risk of developing active tuberculosis (TB). To reduce the burden of TB among people living with HIV (PLHIV), the World Health Organization (WHO) recommends systematic TB screening followed by 1) confirmatory TB testing for all those who screen positive and 2) TB preventive therapy (TPT) for all TPT-eligible PLHIV who screen negative.

The objective of the TB Screening Improves Preventive Therapy Uptake (TB SCRIPT) trial is to determine whether TB screening based on C-reactive protein (CRP) levels, measured using a rapid and low-cost point-of-care (POC) assay, improves TPT uptake and clinical outcomes of PLHIV, relative to symptom-based TB screening.

DETAILED DESCRIPTION:
The overall objective of the TB SCRIPT trial is to evaluate the effectiveness and cost-effectiveness of POC CRP-based TB screening, which is the next step required for successful scale-up of both systematic TB screening and TPT. The study's central hypothesis is that compared to symptom-based TB screening, a TB screening strategy based on CRP levels measured at the point-of-care will improve TPT uptake, thereby reducing TB incidence and its associated mortality among PLHIV.

To test this hypothesis, the investigators will conduct an individual randomized control trial enrolling PLHIV presenting to clinics in Uganda for routine antiretroviral therapy (ART) initiation. Eligible participants will be randomized to either POC CRP-based TB screening (intervention arm) or symptom-based TB screening (control arm). In both arms, screen-positive participants will undergo confirmatory TB testing; participants found to have prevalent TB will be initiated on standard TB treatment. In both arms, screen-negative participants will be assessed for TPT eligibility; TPT-eligible participants will be initiated on standard TPT. All participants will be followed for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Confirmed HIV+ test result
* CD4 T lymphocyte count of ≤ 350 cells/μL
* Capacity to provide written (or witnessed verbal, if illiterate) informed consent

Exclusion Criteria:

* Completed treatment for active pulmonary or extra-pulmonary TB within the past 2 years
* Completed a full course of TPT within the past year
* Actively taking any internationally-approved medication for TB treatment for any reason, within 2 weeks of study entry
* Prior history of combined ART for HIV treatment for any duration (does not include single-dose ART for prevention of vertical transmission of HIV)
* Currently resides 25 km outside their enrollment site, plans to move 25 km outside their enrollment site in the next 2 years, or plans to transfer their HIV care from their current enrollment site

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1719 (Actual)
Dates: Start 2020-11-16 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Microbiologically-confirmed incident TB and all-cause mortality | two years
  Time to first diagnosis of microbiologically-confirmed incident TB or death from any cause

SECONDARY OUTCOMES:
TB incidence: number diagnosed | two years
  Number diagnosed with microbiologically-confirmed incident TB
TB incidence: incidence | two years
  Incidence of microbiologically-confirmed TB (excluding prevalent TB cases)
TB incidence: Time to microbiologically-confirmed incident TB diagnosis | two years
  Days from three months post-enrollment to incident TB diagnosis (or censoring)
TB incidence: incidence rate | two years
  Incident rate of microbiologically-confirmed TB
TB incidence: drug resistant TB | two years
  Number diagnosed with drug-resistant incident TB
TB incidence: drug resistant TB among people receiving TPT | two years
  Proportion of participants receiving TPT diagnosed with incident drug resistant TB
Mortality: number of deaths from any cause | two years
  Number who died from any cause
Mortality: time to death from any cause | two years
  Number of days from enrollment to death from any cause
Mortality: all-cause death rate | two years
  Rate of deaths from any cause
Mortality: number who died from TB | two years
  Number who died from confirmed or probable TB
TPT uptake: number screen-negatives prescribed TPT | two years
  Number of screen-negatives prescribed TPT
TPT uptake: number screen-positives prescribed TPT | two years
  Number screen-positives prescribed TPT
TPT uptake: number initiated on TPT | two years
  Number screen-negatives prescribed TPT + number screen-positives prescribed TPT
TPT uptake: time to TPT initiation | two years
  Days from baseline TB screening to initiation of TPT
TPT uptake: number completing TPT | two years
  Number initiated on TPT who completed ≥90% of treatment over prescribed TPT period
Prevalent TB diagnosis: number microbiologically-confirmed prevalent TB cases detected by screening test | two years
  Number screen-positives diagnosed with prevalent TB
Prevalent TB diagnosis: number microbiologically-confirmed prevalent TB cases missed by screening test | two years
  Number screen-negatives diagnosed with prevalent TB
Prevalent TB diagnosis: number diagnosed with microbiologically-confirmed prevalent TB | two years
  Number screen-positives diagnosed with prevalent TB + number screen-negatives diagnosed with prevalent TB
Prevalent TB treatment: Number treated for prevalent TB | two years
  Number initiated on TB treatment 3 months or less after study entry
Prevalent TB treatment: number with microbiologically-confirmed prevalent TB completing treatment | two years
  Number diagnosed and treated who completed treatment
Prevalent TB treatment: time to treatment of microbiologically-confirmed prevalent TB | two years
  Days from prevalent TB diagnosis to initiation of TB treatment

CONTACTS AND LOCATIONS:
Overall Officials: Christina Yoon, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- Kampala Capital City Authority Clinic, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] WHO. Global Tuberculosis Report 2017. Geneva, Switzerland. World Health Organization 2017.
- [Background] Durovni B, Saraceni V, Moulton LH, Pacheco AG, Cavalcante SC, King BS, Cohn S, Efron A, Chaisson RE, Golub JE. Effect of improved tuberculosis screening and isoniazid preventive therapy on incidence of tuberculosis and death in patients with HIV in clinics in Rio de Janeiro, Brazil: a stepped wedge, cluster-randomised trial. Lancet Infect Dis. 2013 Oct;13(10):852-8. doi: 10.1016/S1473-3099(13)70187-7. Epub 2013 Aug 16. PMID 23954450
- [Background] TEMPRANO ANRS 12136 Study Group; Danel C, Moh R, Gabillard D, Badje A, Le Carrou J, Ouassa T, Ouattara E, Anzian A, Ntakpe JB, Minga A, Kouame GM, Bouhoussou F, Emieme A, Kouame A, Inwoley A, Toni TD, Ahiboh H, Kabran M, Rabe C, Sidibe B, Nzunetu G, Konan R, Gnokoro J, Gouesse P, Messou E, Dohoun L, Kamagate S, Yao A, Amon S, Kouame AB, Koua A, Kouame E, Ndri Y, Ba-Gomis O, Daligou M, Ackoundze S, Hawerlander D, Ani A, Dembele F, Kone F, Guehi C, Kanga C, Koule S, Seri J, Oyebi M, Mbakop N, Makaila O, Babatunde C, Babatounde N, Bleoue G, Tchoutedjem M, Kouadio AC, Sena G, Yededji SY, Assi R, Bakayoko A, Mahassadi A, Attia A, Oussou A, Mobio M, Bamba D, Koman M, Horo A, Deschamps N, Chenal H, Sassan-Morokro M, Konate S, Aka K, Aoussi E, Journot V, Nchot C, Karcher S, Chaix ML, Rouzioux C, Sow PS, Perronne C, Girard PM, Menan H, Bissagnene E, Kadio A, Ettiegne-Traore V, Moh-Semde C, Kouame A, Massumbuko JM, Chene G, Dosso M, Domoua SK, N'Dri-Yoman T, Salamon R, Eholie SP, Anglaret X. A Trial of Early Antiretrovirals and Isoniazid Preventive Therapy in Africa. N Engl J Med. 2015 Aug 27;373(9):808-22. doi: 10.1056/NEJMoa1507198. Epub 2015 Jul 20. PMID 26193126
- [Background] Rangaka MX, Wilkinson RJ, Boulle A, Glynn JR, Fielding K, van Cutsem G, Wilkinson KA, Goliath R, Mathee S, Goemaere E, Maartens G. Isoniazid plus antiretroviral therapy to prevent tuberculosis: a randomised double-blind, placebo-controlled trial. Lancet. 2014 Aug 23;384(9944):682-90. doi: 10.1016/S0140-6736(14)60162-8. Epub 2014 May 13. PMID 24835842
- [Background] Grant AD, Charalambous S, Fielding KL, Day JH, Corbett EL, Chaisson RE, De Cock KM, Hayes RJ, Churchyard GJ. Effect of routine isoniazid preventive therapy on tuberculosis incidence among HIV-infected men in South Africa: a novel randomized incremental recruitment study. JAMA. 2005 Jun 8;293(22):2719-25. doi: 10.1001/jama.293.22.2719. PMID 15941800
- [Background] Churchyard GJ, Fielding KL, Lewis JJ, Coetzee L, Corbett EL, Godfrey-Faussett P, Hayes RJ, Chaisson RE, Grant AD; Thibela TB Study Team. A trial of mass isoniazid preventive therapy for tuberculosis control. N Engl J Med. 2014 Jan 23;370(4):301-10. doi: 10.1056/NEJMoa1214289. PMID 24450889
- [Background] WHO. Guidelines for intensified tuberculosis case-finding and isoniazid preventive therapy for people living with HIV in resource-constrained settings. Geneva, Switzerland. World Health Organization 2011.
- [Background] Latent tuberculosis infection: updated and consolidated guidelines for programmatic management [Internet]. Geneva: World Health Organization; 2018. Available from http://www.ncbi.nlm.nih.gov/books/NBK531235/ PMID 30277688
- [Background] Getahun H, Kittikraisak W, Heilig CM, Corbett EL, Ayles H, Cain KP, Grant AD, Churchyard GJ, Kimerling M, Shah S, Lawn SD, Wood R, Maartens G, Granich R, Date AA, Varma JK. Development of a standardized screening rule for tuberculosis in people living with HIV in resource-constrained settings: individual participant data meta-analysis of observational studies. PLoS Med. 2011 Jan 18;8(1):e1000391. doi: 10.1371/journal.pmed.1000391. PMID 21267059
- [Background] WHO. High-priority target product profiles for new tuberculosis diagnostics: report of a consensus meeting. Geneva, Switzerland. World Health Organization 2014.
- [Background] Lawn SD, Brooks SV, Kranzer K, Nicol MP, Whitelaw A, Vogt M, Bekker LG, Wood R. Screening for HIV-associated tuberculosis and rifampicin resistance before antiretroviral therapy using the Xpert MTB/RIF assay: a prospective study. PLoS Med. 2011 Jul;8(7):e1001067. doi: 10.1371/journal.pmed.1001067. Epub 2011 Jul 26. PMID 21818180
- [Background] Kufa T, Mngomezulu V, Charalambous S, Hanifa Y, Fielding K, Grant AD, Wada N, Chaisson RE, Churchyard GJ, Gounder CR. Undiagnosed tuberculosis among HIV clinic attendees: association with antiretroviral therapy and implications for intensified case finding, isoniazid preventive therapy, and infection control. J Acquir Immune Defic Syndr. 2012 Jun 1;60(2):e22-8. doi: 10.1097/QAI.0b013e318251ae0b. PMID 22627184
- [Background] Swindells S, Komarow L, Tripathy S, Cain KP, MacGregor RR, Achkar JM, Gupta A, Veloso VG, Asmelash A, Omoz-Oarhe AE, Gengiah S, Lalloo U, Allen R, Shiboski C, Andersen J, Qasba SS, Katzenstein DK; AIDS Clinical Trials Group 5253 Study Team. Screening for pulmonary tuberculosis in HIV-infected individuals: AIDS Clinical Trials Group Protocol A5253. Int J Tuberc Lung Dis. 2013 Apr;17(4):532-9. doi: 10.5588/ijtld.12.0737. PMID 23485388
- [Background] Henostroza G, Harris JB, Chitambi R, Siyambango M, Turnbull ER, Maggard KR, Kruuner A, Kapata N, Reid SE. High prevalence of tuberculosis in newly enrolled HIV patients in Zambia: need for enhanced screening approach. Int J Tuberc Lung Dis. 2016 Aug;20(8):1033-9. doi: 10.5588/ijtld.15.0651. PMID 27393536
- [Background] DERBES VJ, JACOBS S, LINN RH, TURNER M, WALSH JJ. C-reactive protein in pulmonary tuberculosis. Am Rev Tuberc. 1956 Sep;74(3):464-7. doi: 10.1164/artpd.1956.74.3.464. No abstract available. PMID 13354933
- [Background] Ganter U, Arcone R, Toniatti C, Morrone G, Ciliberto G. Dual control of C-reactive protein gene expression by interleukin-1 and interleukin-6. EMBO J. 1989 Dec 1;8(12):3773-9. doi: 10.1002/j.1460-2075.1989.tb08554.x. PMID 2555173
- [Background] Ogawa T, Uchida H, Kusumoto Y, Mori Y, Yamamura Y, Hamada S. Increase in tumor necrosis factor alpha- and interleukin-6-secreting cells in peripheral blood mononuclear cells from subjects infected with Mycobacterium tuberculosis. Infect Immun. 1991 Sep;59(9):3021-5. doi: 10.1128/iai.59.9.3021-3025.1991. PMID 1879927
- [Background] Saunders R, Robson S, Soule S, Kirsch RE. Secretion of interleukin-6 by peripheral blood mononuclear cells from patients with pulmonary tuberculosis and their contacts. J Clin Lab Immunol. 1993;40(1):19-28. PMID 7932624
- [Background] Flesch IE, Kaufmann SH. Role of cytokines in tuberculosis. Immunobiology. 1993 Nov;189(3-4):316-39. doi: 10.1016/S0171-2985(11)80364-5. PMID 8125515
- [Background] Weinhold B, Ruther U. Interleukin-6-dependent and -independent regulation of the human C-reactive protein gene. Biochem J. 1997 Oct 15;327 ( Pt 2)(Pt 2):425-9. doi: 10.1042/bj3270425. PMID 9359411
- [Background] Gabay C, Kushner I. Acute-phase proteins and other systemic responses to inflammation. N Engl J Med. 1999 Feb 11;340(6):448-54. doi: 10.1056/NEJM199902113400607. No abstract available. PMID 9971870
- [Background] Lawn SD, Wiktor S, Coulibaly D, Ackah AN, Lal RB. Serum C-reactive protein and detection of tuberculosis in persons co-infected with the human immunodeficiency virus. Trans R Soc Trop Med Hyg. 2001 Jan-Feb;95(1):41-2. doi: 10.1016/s0035-9203(01)90328-1. No abstract available. PMID 11280064
- [Background] Kihara M, Kamakura M, Feldman MD. Introduction: HIV/AIDS surveillance in a new era. J Acquir Immune Defic Syndr. 2003 Feb;32 Suppl 1:S1-2. doi: 10.1097/00126334-200302011-00001. No abstract available. PMID 12571508
- [Background] Drain PK, Kupka R, Msamanga GI, Urassa W, Mugusi F, Fawzi WW. C-reactive protein independently predicts HIV-related outcomes among women and children in a resource-poor setting. AIDS. 2007 Oct 1;21(15):2067-75. doi: 10.1097/QAD.0b013e32826fb6c7. PMID 17885297
- [Background] Kuller LH, Tracy R, Belloso W, De Wit S, Drummond F, Lane HC, Ledergerber B, Lundgren J, Neuhaus J, Nixon D, Paton NI, Neaton JD; INSIGHT SMART Study Group. Inflammatory and coagulation biomarkers and mortality in patients with HIV infection. PLoS Med. 2008 Oct 21;5(10):e203. doi: 10.1371/journal.pmed.0050203. PMID 18942885
- [Background] Tien PC, Schneider MF, Cox C, Cohen M, Karim R, Lazar J, Young M, Glesby MJ. HIV, HAART, and lipoprotein particle concentrations in the Women's Interagency HIV Study. AIDS. 2010 Nov 27;24(18):2809-17. doi: 10.1097/QAD.0b013e32833fcb3b. PMID 20871387
- [Background] Neuhaus J, Jacobs DR Jr, Baker JV, Calmy A, Duprez D, La Rosa A, Kuller LH, Pett SL, Ristola M, Ross MJ, Shlipak MG, Tracy R, Neaton JD. Markers of inflammation, coagulation, and renal function are elevated in adults with HIV infection. J Infect Dis. 2010 Jun 15;201(12):1788-95. doi: 10.1086/652749. PMID 20446848
- [Background] Shikuma CM, Ribaudo HJ, Zheng Y, Gulick RM, Meyer WA, Tashima KT, Bastow B, Kuritzkes DR, Glesby MJ; AIDS Clinical Trials Group A5095 Study Team. Change in high-sensitivity c-reactive protein levels following initiation of efavirenz-based antiretroviral regimens in HIV-infected individuals. AIDS Res Hum Retroviruses. 2011 May;27(5):461-8. doi: 10.1089/aid.2010.0154. Epub 2010 Nov 23. PMID 20863238
- [Background] Lawn SD, Obeng J, Acheampong JW, Griffin GE. Resolution of the acute-phase response in West African patients receiving treatment for pulmonary tuberculosis. Int J Tuberc Lung Dis. 2000 Apr;4(4):340-4. PMID 10777083
- [Background] Polzin A, Pletz M, Erbes R, Raffenberg M, Mauch H, Wagner S, Arndt G, Lode H. Procalcitonin as a diagnostic tool in lower respiratory tract infections and tuberculosis. Eur Respir J. 2003 Jun;21(6):939-43. doi: 10.1183/09031936.03.00055103. PMID 12797485
- [Background] Schleicher GK, Herbert V, Brink A, Martin S, Maraj R, Galpin JS, Feldman C. Procalcitonin and C-reactive protein levels in HIV-positive subjects with tuberculosis and pneumonia. Eur Respir J. 2005 Apr;25(4):688-92. doi: 10.1183/09031936.05.00067604. PMID 15802344
- [Background] Choi CM, Kang CI, Jeung WK, Kim DH, Lee CH, Yim JJ. Role of the C-reactive protein for the diagnosis of TB among military personnel in South Korea. Int J Tuberc Lung Dis. 2007 Feb;11(2):233-6. PMID 17263297
- [Background] Breen RA, Leonard O, Perrin FM, Smith CJ, Bhagani S, Cropley I, Lipman MC. How good are systemic symptoms and blood inflammatory markers at detecting individuals with tuberculosis? Int J Tuberc Lung Dis. 2008 Jan;12(1):44-9. PMID 18173876
- [Background] Kang YA, Kwon SY, Yoon HI, Lee JH, Lee CT. Role of C-reactive protein and procalcitonin in differentiation of tuberculosis from bacterial community acquired pneumonia. Korean J Intern Med. 2009 Dec;24(4):337-42. doi: 10.3904/kjim.2009.24.4.337. Epub 2009 Nov 27. PMID 19949732
- [Background] Sage EK, Noursadeghi M, Evans HE, Parker SJ, Copas AJ, Edwards SG, Miller RF. Prognostic value of C-reactive protein in HIV-infected patients with Pneumocystis jirovecii pneumonia. Int J STD AIDS. 2010 Apr;21(4):288-92. doi: 10.1258/ijsa.2010.009551. PMID 20378904
- [Background] Wilson D, Badri M, Maartens G. Performance of serum C-reactive protein as a screening test for smear-negative tuberculosis in an ambulatory high HIV prevalence population. PLoS One. 2011 Jan 10;6(1):e15248. doi: 10.1371/journal.pone.0015248. PMID 21249220
- [Background] Lawn SD, Kerkhoff AD, Vogt M, Wood R. Diagnostic and prognostic value of serum C-reactive protein for screening for HIV-associated tuberculosis. Int J Tuberc Lung Dis. 2013 May;17(5):636-43. doi: 10.5588/ijtld.12.0811. PMID 23575330
- [Background] Yoon C, Davis JL, Huang L, Muzoora C, Byakwaga H, Scibetta C, Bangsberg DR, Nahid P, Semitala FC, Hunt PW, Martin JN, Cattamanchi A. Point-of-care C-reactive protein testing to facilitate implementation of isoniazid preventive therapy for people living with HIV. J Acquir Immune Defic Syndr. 2014 Apr 15;65(5):551-6. doi: 10.1097/QAI.0000000000000085. PMID 24346636
- [Background] Yoon C, Chaisson LH, Patel SM, Allen IE, Drain PK, Wilson D, Cattamanchi A. Diagnostic accuracy of C-reactive protein for active pulmonary tuberculosis: a meta-analysis. Int J Tuberc Lung Dis. 2017 Sep 1;21(9):1013-1019. doi: 10.5588/ijtld.17.0078. PMID 28826451
- [Background] Shapiro AE, Hong T, Govere S, Thulare H, Moosa MY, Dorasamy A, Wallis CL, Celum CL, Grosset J, Drain PK. C-reactive protein as a screening test for HIV-associated pulmonary tuberculosis prior to antiretroviral therapy in South Africa. AIDS. 2018 Aug 24;32(13):1811-1820. doi: 10.1097/QAD.0000000000001902. PMID 29847333
- [Background] Yoon C, Semitala FC, Atuhumuza E, Katende J, Mwebe S, Asege L, Armstrong DT, Andama AO, Dowdy DW, Davis JL, Huang L, Kamya M, Cattamanchi A. Point-of-care C-reactive protein-based tuberculosis screening for people living with HIV: a diagnostic accuracy study. Lancet Infect Dis. 2017 Dec;17(12):1285-1292. doi: 10.1016/S1473-3099(17)30488-7. Epub 2017 Aug 25. PMID 28847636
- [Background] Yoon C, Semitala FC, Asege L, Katende J, Mwebe S, Andama AO, Atuhumuza E, Nakaye M, Armstrong DT, Dowdy DW, McCulloch CE, Kamya M, Cattamanchi A. Yield and Efficiency of Novel Intensified Tuberculosis Case-Finding Algorithms for People Living with HIV. Am J Respir Crit Care Med. 2019 Mar 1;199(5):643-650. doi: 10.1164/rccm.201803-0490OC. PMID 30192649
- [Background] Rajan JV, Semitala FC, Mehta T, Seielstad M, Montalvo L, Andama A, Asege L, Nakaye M, Katende J, Mwebe S, Kamya MR, Yoon C, Cattamanchi A. A Novel, 5-Transcript, Whole-blood Gene-expression Signature for Tuberculosis Screening Among People Living With Human Immunodeficiency Virus. Clin Infect Dis. 2019 Jun 18;69(1):77-83. doi: 10.1093/cid/ciy835. PMID 30462176
- [Background] Chaisson LH, Semitala FC, Asege L, Mwebe S, Katende J, Nakaye M, Andama AO, Marquez C, Atuhumuza E, Kamya M, Cattamanchi A, Yoon C. Point-of-care C-reactive protein and risk of early mortality among adults initiating antiretroviral therapy. AIDS. 2019 Apr 1;33(5):895-902. doi: 10.1097/QAD.0000000000002130. PMID 30649057
- [Background] Semitala FC, Cattamanchi A, Andama A, Atuhumuza E, Katende J, Mwebe S, Asege L, Nakaye M, Kamya MR, Yoon C. Brief Report: Yield and Efficiency of Intensified Tuberculosis Case-Finding Algorithms in 2 High-Risk HIV Subgroups in Uganda. J Acquir Immune Defic Syndr. 2019 Dec 1;82(4):416-420. doi: 10.1097/QAI.0000000000002162. PMID 31658185
- [Background] Uganda Ministry of Health. Report on the Population-based survey of prevalence of tuberculosis disease in Uganda 2014-2015. Kampala: MOH, 2017.
- [Background] PEPFAR Uganda Program data. (https://www.pepfar.gov/documents/organization/285851.)
- [Background] Yung-Pin C. Biased coin design with imbalance tolerance. Stochastic Models. 1999 Jan 1;15(5):953-75. doi: 10.1080/15326349908807570
- [Background] Pfafflin A, Schleicher E. Inflammation markers in point-of-care testing (POCT). Anal Bioanal Chem. 2009 Mar;393(5):1473-80. doi: 10.1007/s00216-008-2561-3. Epub 2008 Dec 23. PMID 19104782
- [Background] Claus DR, Osmand AP, Gewurz H. Radioimmunoassay of human C-reactive protein and levels in normal sera. J Lab Clin Med. 1976 Jan;87(1):120-8. PMID 1245780
- [Background] Gupta A, Montepiedra G, Aaron L, Theron G, McCarthy K, Bradford S, Chipato T, Vhembo T, Stranix-Chibanda L, Onyango-Makumbi C, Masheto GR, Violari A, Mmbaga BT, Aurpibul L, Bhosale R, Mave V, Rouzier V, Hesseling A, Shin K, Zimmer B, Costello D, Sterling TR, Chakhtoura N, Jean-Philippe P, Weinberg A; IMPAACT P1078 TB APPRISE Study Team. Isoniazid Preventive Therapy in HIV-Infected Pregnant and Postpartum Women. N Engl J Med. 2019 Oct 3;381(14):1333-1346. doi: 10.1056/NEJMoa1813060. PMID 31577875
- [Background] Uganda Ministry of Health. Isoniazid preventive therapy in Uganda: a health worker's guide. Kampala: MOH, 2014.
- [Derived] Semitala FC, Chaisson LH, Dowdy DW, Armstrong DT, Opira B, Aman K, Kamya M, Phillips PPJ, Yoon C. Tuberculosis screening improves preventive therapy uptake (TB SCRIPT) trial among people living with HIV in Uganda: a study protocol of an individual randomized controlled trial. Trials. 2022 May 12;23(1):399. doi: 10.1186/s13063-022-06371-0. PMID 35550621